CLINICAL TRIAL: NCT06058884
Title: Predictors of the Unfavourable Outcomes in Acute Ischemic Stroke Patients Treated With Alteplase, a Multi-centre Prospective Study
Brief Title: Predictors of AIS Unfavorable Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, Dr., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23091988
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Ischemic Stroke; Alteplase Adverse Reaction
Keywords: alteplase; acute ischemic stroke; Egypt; Saudi Arabia
MeSH Terms: conditions — Ischemic Stroke | interventions — Tissue Plasminogen Activator

STUDY DESIGN:
Intervention Model Description: The study consisted of two distinct groups. The first group consisted of 456 patients who experienced favourable outcomes (mRS two or less), while the second group comprised 136 patients who experienced unfavourable outcomes (mRS more than two).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- favourbale outcome group (Active Comparator): Four hundred fifty-six acute ischemic stroke (AIS) patients who had modified Rankin scale (mRS) two or less after 90 days of ischemic stroke.
  Interventions: Drug: Alteplase
- unfavourbale outcome group (Active Comparator): One hundred thirty-six acute ischemic stroke (AIS) patients who had modified Rankin scale (mRS) three or more after 90 days of ischemic stroke.
  Interventions: Drug: Alteplase

INTERVENTIONS:
Drug: Alteplase — Following the guidelines set forth by the American Heart Association/American Stroke Association (AHA/ASA), inclusion and exclusion criteria for alteplase were established; 0.9 mg/kg of alteplase up to a maximum dose of 90 mg was administered intravenously to eligible individuals within 4.5 hours of the beginning of their clinical manifestations (10% bolus, 90% infusion in 1 hour). After receiving IV-alteplase, all patients continued their management and rehabilitation in the stroke unit.

SUMMARY:
The investigators evaluated whether the characteristics of ischemic stroke patients, door-to-needle time, and stroke risk factors were predictive variables for unfavourable outcomes.

DETAILED DESCRIPTION:
Investigators conducted a prospective cohort study between January 2022 and June 2023 and screened 1184 patients presented with AIS and received alteplase and included 592 AIS patients who met the inclusion criteria and were diagnosed based on a thorough clinical assessment, including a detailed medical history, physical examination and specific brain imaging results and treated with alteplase within four and half hours of stroke onset.

The investigators assessed mRS after 90 days via a 10-minute telephone interview. With patients or their primary caregivers to detect the score, all of our patients had baseline mRS of zero. mRS two or less was considered a favourable outcome

The study consisted of two distinct groups. The first group consisted of 456 patients who experienced favourable outcomes, while the second group comprised 136 patients who experienced unfavourable outcomes.

The investigators evaluated whether the characteristics of ischemic stroke patients, door-to-needle time, and stroke risk factors were predictive variables for unfavourable outcomes.

ELIGIBILITY:
Inclusion Criteria:

The investigators enrolled individuals of both genders, aged between 18 and 75, who presented with acute first-ever ischemic stroke and were eligible for thrombolysis.

Exclusion Criteria:

* The investigators excluded patients who had not been followed up on for 90 days after enrollment,
* Those with alteplase contraindications or did not receive the total dose of alteplase due to any reason were excluded
* The investigators excluded patients with a known history of persistent or recurrent CNS pathology (e.g., epilepsy, meningioma, multiple sclerosis, history of head trauma with a residual neurological deficit).
* The investigators excluded patients who had recurrent ischemic stroke diagnosed by appropriate clinical history and/or MRI brain findings.
* The investigators excluded patients with symptoms of major organ failure, active malignancies, or an acute myocardial infarction within the previous six weeks.
* The investigators also excluded pregnant and lactating patients with stroke due to venous thrombosis and stroke following cardiac arrest.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
modified Rankin scale (mRS) | 90 days
  To detect the score, investigators assessed modified rankin scale (mRS) after 90 days via a 10-minute telephone interview with patients or their primary caregivers. mRS two or less was considered a favourable outcome.
  mRS is a scale that assessed the outcome of stroke patients and its score ranged from zero to six. the lower the values the better the outcome
predictors of the unfavourable outcomes | 90 days
  The investigators employed univariate and multivariate Logistic regression analysis to assess the ability of patients' characteristics and risk factors to predict the unfavourable outcomes after 90 days of acute ischemic stroke.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD,PHD, Principal Investigator — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data supporting this research's findings may be available from the principal investigator, Mohamed G. Zeinhom, upon reasonable request.

REFERENCES:
- [Result] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Result] Zeinhom MG, Aref HM, El-Khawas H, Roushdy TM, Shokri HM, Elbassiouny A. A pilot study of the ticagrelor role in ischemic stroke secondary prevention. Eur Neurol. 2022;85(1):50-55. doi: 10.1159/000518786. Epub 2021 Aug 30. PMID 34515113
- [Result] Bruno A, Levine SR, Frankel MR, Brott TG, Lin Y, Tilley BC, Lyden PD, Broderick JP, Kwiatkowski TG, Fineberg SE; NINDS rt-PA Stroke Study Group. Admission glucose level and clinical outcomes in the NINDS rt-PA Stroke Trial. Neurology. 2002 Sep 10;59(5):669-74. doi: 10.1212/wnl.59.5.669. PMID 12221155
- [Result] Aref HM, El-Khawas H, Elbassiouny A, Shokri HM, Zeinhom MG, Roushdy TM. A randomized pilot study of the efficacy and safety of loading ticagrelor in acute ischemic stroke. Neurol Sci. 2023 Feb;44(2):765-771. doi: 10.1007/s10072-022-06525-7. Epub 2022 Nov 30. PMID 36446950
- [Result] Ahmed SR, Mohamed AAM, Salem HH, Helmy S, Moustafa RR, Borham SMF. Association of white matter hyperintensities with migraine phenotypes and response to treatment. Acta Neurol Belg. 2023 Oct;123(5):1725-1733. doi: 10.1007/s13760-022-02015-x. Epub 2022 Jul 19. PMID 35854172
- [Derived] Zeinhom MG, Khalil MFE, Kamel IFM, Kohail AM, Ahmed SR, Elbassiouny A, Shuaib A, Al-Nozha OM. Predictors of the unfavorable outcomes in acute ischemic stroke patients treated with alteplase, a multi-center randomized trial. Sci Rep. 2024 Mar 12;14(1):5960. doi: 10.1038/s41598-024-56067-5. PMID 38472241